CLINICAL TRIAL: NCT05136508
Title: The Effect of Volatile Anesthesia and Total Intravenous Anesthesia on Shedding of the Endothelial Glycocalyx in Patients Undergoing Mastectomy and Breast Reconstruction Using Deep Inferior Epigastric Artery Perforator Free Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2021-0401
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Deep Inferior Epigastric Artery Perforator Flap Breast Reconstruction
Keywords: syndecan-1; propofol; volatile; anesthesia; deep inferior epigastric artery perforator flap breast reconstruction
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA (Experimental): In the TIVA group, anesthesia was induced with TCI of propofol (Ce of 4.0-4.5 μg/ml) and remifentanil (Ce of 4.0 ng/ml). Anesthesia was maintained with TCI of propofol and remifentanil. Anesthesia depth was adjusted to maintain a PSI of 25-50.
  Interventions: Drug: Propofol
- Inhalation (Active Comparator): In the volatile group, anesthesia was induced with an intravenous bolus of propofol 1.0-1.5 mg/kg and TCI of remifentanil (effect-site concentration [Ce] of 4.0 ng/ml). Anesthesia was maintained with sevoflurane (0.8-1 age-adjusted minimum alveolar concentration) and TCI of remifentanil
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Anesthesia was induced with TCI of propofol (Ce of 4.0-4.5 μg/ml) and remifentanil (Ce of 4.0 ng/ml). Anesthesia was maintained with TCI of propofol and remifentanil. Anesthesia depth was adjusted to maintain a PSI of 25-50.
  Other Names: TIVA group
  Arms: TIVA
Drug: Sevoflurane — Anesthesia was induced with an intravenous bolus of propofol 1.5-2 mg/kg and TCI of remifentanil (effect-site concentration [Ce] of 4.0 ng/ml). Anesthesia was maintained with sevoflurane (0.8-1 age-adjusted minimum alveolar concentration) and TCI of remifentanil
  Other Names: volatile group
  Arms: Inhalation

SUMMARY:
The aim of this study was to investigate the effects of total intravenous and inhalation anesthesia on the damage of endothelial glucocorticoids by comparing the concentration of syndecan-1 in patients undergoing mastectomy and breast reconstruction using deep inferior epigastric artery perforator free flap

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of total intravenous and inhalation anesthesia on the damage of endothelial glucocorticoids by comparing the concentration of syndecan-1 in patients undergoing mastectomy and breast reconstruction using deep inferior epigastric artery perforator free flap

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 20 years old with ASA class I-III
2. Scheduled total mastectomy and deep inferior epigastric artery perforator flap breast reconstruction

Exclusion Criteria:

1. emergency surgery
2. Bilateral deep inferior epigastric artery perforator flap breast reconstruction
3. patients unable to make their own decisions, illiterate, foreigners
4. Allergy / hypersensitivity to sevoflurane or propofol 5, Current or past history or thrombosis / thromboembolism

6. patients who are taking oral contraceptives 7. Patients with renal insufficiency (eGFR 60 ml / min / 1.73 m 2 or less) 8. Patients receiving anticoagulants 9. pregnant and lactating women 10. Patients with history of psychiatric disease or neurological disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Changes in blood concentration of syndecan-1 | 1) 10 minutes after anesthesia induction <before surgery(base concentration)> 2) 10 minutes after sitting position 3) 1 hour after surgery
  Blood levels of syndecan-1 are assessed at 10 minutes after anesthesia induction, 10 minutes after sitting position, and 1 hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided